CLINICAL TRIAL: NCT02693236
Title: Clinical Research of Genetically Modified Dendritic Cells in Combination With Cytokine-induced Killer Cell Treatment in Middle and Advanced Esophagus Cancer Patients
Brief Title: DC Vaccine Combined With CIK Cells in Patients With Esophagus Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-DC/CIK-EC
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2015-10

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenovirus-transfected autologous DC vaccine plus CIK cells (Experimental)
  Interventions: Biological: adenovirus-transfected autologous DC vaccine plus CIK cells

INTERVENTIONS:
Biological: adenovirus-transfected autologous DC vaccine plus CIK cells

SUMMARY:
The aim of this Phase I/II study is to evaluate the safety and efficacy of dendritic cells(DC) combined with cytokine-induced killer (CIK) cells in patients with advanced esophagus cancer. Experimental recombinant adenovirus coded mRNA including MUC1 and Survivin that transfected DC, which are used for DC-based immunotherapy. Based on the results of our previously performed preclinical study with DC vaccine combined with CIK cells, the researcher plan to perform the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of esophagus cancer
* Age >18 years at time of consent
* Received standardized treatment of Small-Cell Lung Cancer
* Interval between the last standardized treatment and DC/CIK treatment ≥ 4weeks
* KPS (Karnofsky performance scale) >60
* Patient's written informed consent
* No severe viral or bacterial infections
* Predicted survival >3 months

Exclusion Criteria:

* Serious dysfunction of vital organs(heart, liver or kidney)
* History of autoimmune diseases
* Pregnant and breast-feeding patient
* Active or chronic infectious diseases
* History of allergy or hypersensitivity to study product excipients
* Currently participating in another clinical trial
* Received chemotherapy, radiotherapy, immune inhibitor (such as corticosteroid) or other immunotherapy (such as vaccine) during prior 4 weeks
* Clinically relevant diseases or infections (HBV, HCV, HIV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
objective rate response (CR+PR) as measured by RECIST criteria | Time Frame: 4 weeks after DC/CIK treatment

SECONDARY OUTCOMES:
number of participants with adverse events | Time Frame: 3 days within DC/CIK treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes